CLINICAL TRIAL: NCT04521218
Title: Comparison of Thrust Joint Manipulation and Reverse SNAGS (Sustained Natural Apophyseal Glides) of Upper Cervical Spine in Cervicogenic Headache
Brief Title: Thrust Joint Manipulation and Reverse SNAGS (Sustained Natural Apophyseal Glides) in Cervicogenic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00694 Amna Arshad
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cervicogenic Headache
Keywords: Thrust joint manipulation; Reverse sustained natural apophyseal glides; Cervicogenic headache; Mobilization and Manipulation
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thrust joint Manipulation (Experimental): Thrust joint Manipulation, heat application, Strengthening exercise and home plan
  Interventions: Other: Thrust Joint Manipulation
- Reverse Sustained Natural apophyseal glides (Active Comparator): Reverse Sustained Natural apophyseal glides (SNAG), heat application, Strengthening exercise and home plan.
  Interventions: Other: Reverse Sustained Natural apophyseal glides

INTERVENTIONS:
Other: Thrust Joint Manipulation — Experimental group included TJM, Cervical hot pack, strengthening exercises and home plan; 3 sessions of manipulation per week and total of 4 weeks. Measurement will be taken at base level and after the last session, i.e. Pain intensity, pain pressure threshold, ROM, and disability.
  These exercises included. Cervical Flexion, Extension Rotation, lateral flexion and back strengthening exercises. These all exercises were performed 3 x 15 Repetitions with 10 sec hold. This protocol was for 4 weeks and 3 sessions per week.
  Home plan exercises includes Craniocervical Flexion, Craniocervical Extension, Rotation Exercise, Lateral Flexion Exercise, Chin Tuck in and Shoulder blade exercise were advised to perform 3 x 10 Repetition with 10 - 30 sec hold.
  Arms: Thrust joint Manipulation
Other: Reverse Sustained Natural apophyseal glides — Control group included Moist Hot Pack (Cervical contour- 8.25 x 10 x 2) for 10 Mins, Reverse SNAGS (10 Repetitions holding for 10 sec in each glide with a rest time of 30 seconds in between), Strengthening exercise and home plan. 3 sessions of mobilization per week and total of 4 weeks. Measurement will be taken at base level and after the last session, i.e. Pain intensity, pain pressure threshold, ROM, and disability.
  These exercises included. Cervical Flexion, Extension Rotation, lateral flexion and back strengthening exercises. These all exercises were performed 3 x 15 Repetitions with 10 sec hold. This protocol was for 4 weeks and 3 sessions per week.
  Home plan exercises includes Craniocervical Flexion, Craniocervical Extension, Rotation Exercise, Lateral Flexion Exercise, Chin Tuck in and Shoulder blade exercise were advised to perform 3 x 10 Repetition with 10 - 30 sec hold
  Arms: Reverse Sustained Natural apophyseal glides

SUMMARY:
The purpose of the study was to compare the effect of upper cervical thrust joint manipulation and reverse Sustained Natural apophyseal Glide on intensity of pain, pain pressure threshold, range of motion and headache disability in patients with cervicogenic headache. A randomized control trial was conducted at Max Rehab and Physical therapy center, Islamabad. The sample size was calculated through open epi tool is 16. The participants were divided in two groups, 8 participants in experimental group and 8 participants in control group. The study duration was six months. Sampling technique applied was Purposive sampling for recruitment and group randomization using sealed envelope method. Only 20 to 40 years participants with cervicogenic headache and associated symptoms were included in the study. Tools used in this study are Numeric pain rating Scale (NPRS), Algometer, Inclinometer and headache disability index (HDI). Data analyzed through Statistical Package for the Social Sciences (SPSS) version 23.

DETAILED DESCRIPTION:
In 1983 the term "cervicogenic headache" was introduced in an article in the medical literature. The diagnostic criteria of cervicogenic headache was revised in 1998. The international headache society classified the types of headaches based on their source and characteristics. Studies showed that out of 47% of the patients suffering from headache. 38% are tension-type ; 10% are migraine ; 3% chronic headache and 2.5 to 4.1 % are cervicogenic headaches.The prevalence of cervicogenic headache (CH) after the whiplash is as high as fifty-three percent.Literature revealed that due to varying use of diagnostic measures it is difficult to find out the true prevalence of cervicogenic headache but it ranges from minimum 0.7% to maximum 13.8% in population.

The headache which is originated from the cervical spine and pain is referred to the head region is termed as Cervicogenic headache.So, the source of pain is a cervical region located near the base of the skull, pain is referred from the neck region which travels towards the occulo-frontal and temporal areas of the head.Cervicogenic headache is four times more prevalent in females than males. Females suffer more from cervicogenic head due to hormonal imbalances and poor posture. Poor posture includes the forward headache posture which affects the normal biomechanics of the cervical spine and increases the stress on the neck region.

The possible cause of cervicogenic headache is said to be the supply of the upper three cervical nerves and its various distributions.Upper three cervical nerves innervate the atlantoaxial joint, atlantooccipital joint, facet joint (C2-C3), suboccipital, paravertebral. upper posterior neck musculature, upper cervical ligaments, spinal dura mater, the vertebral artery, intervertebral disc (C2-C3), trapezius, and sternocleidomastoid muscles. Any of these structures is the possible source of pain and it should be diagnosed first. According to the criteria of the International headache society (IHS) impairment in the function of upper cervical muscles is the source of cervicogenic headache.Patients suffering from cervicogenic headaches show a decrease in their quality of life and also compromised physical abilities as compared to other types of headaches.

A multifaced approach is required to treat the patients suffering from cervicogenic headaches. Most commonly pharmacological, non-pharmacological, physical therapy, anesthetic blockade, and sometimes surgical approach is used. A successful intervention requires a multidisciplinary team of physicians including a pain specialist, anesthesiologist, physical therapist, a psychologist to provide a suitable treatment. For the long-lasting effect of the nerve blocks and neurolytic procedures, physical therapy and rehabilitation are required.

Different physical therapy treatments including thrust joint manipulation, mobilizations, exercise program, postural education, or modification used as an effective intervention of cervicogenic headache. A combination of these treatments is used to subside the symptoms of CH.

Literature review:

A systematic and evidence-based search of relevant literature was performed by utilizing PubMed and Google Scholar as search engines and the key words used were sustained natural apophyseal glides, thrust joint manipulation, mulligan, and reverse sustained natural apophyseal glides. The purpose of the literature review is to find out the pre-existing literature regarding the Reverse SNAGS and TJM interventions for cervicogenic headache.

According to a systematic review and meta-analysis conducted in 2019 on cervicogenic headache to find out the effectiveness of mobilization and manipulation compared to other conservative interventions in reducing pain and disability. So, it was concluded that both mobilization and manipulation are effective in cervicogenic headache but there were few limitations in the study that only nine studies were included and more quality research are required. Further research is required to observe the long-term effect and other interventions for clinical effectiveness.

An overview of systematic reviews was conducted in 2019 on the physical therapy interventions for cervicogenic headache. Results from the reviews stated that manipulation, mobilization, and other conservative interventions were effective in decreasing the frequency of pain and disability in patients suffering from cervicogenic headaches.

According to a randomized control trial conducted in 2019 on cervicogenic headache. The purpose of the study was to determine the effectiveness of headache sustained natural apophyseal glide (SNAG) and SNAG rotation separately as well as in combination in patients suffering from cervicogenic headache to reduce the headache and improve activity limitation. The results of the study showed that group that received both SNAG and SNAG rotation technique is effective in reducing cervicogenic headache.

A randomized control trail in 2018 on cervicogenic headaches. The purpose of the study was to compare the effectiveness of SNAG and reverse SNAG on patients suffering from cervicogenic headache. Results showed that headache SNAG was more effective than reverse SNAG in treating patients suffering from cervicogenic headache. The major limitation of the study was limited sample size and lack of quantitative equipment for measuring the change.

In recent studies, results reported that Sustained Natural Apophyseal Glides and Thrust Joint Manipulation (TJM) were effective in the management of Cervicogenic Headache. However, they did not report if manipulation resulted in superior outcomes compared to mobilization for the management of this population, or secondly no literature was found regarding the reverse SNAGs as an intervention for cervicogenic headache. The purpose of this study is to compare the effects of reverse SNAG and TJM in patients with cervicogenic headache regarding the improvement of headache, pain, pain pressure threshold, and cervical range of motion

ELIGIBILITY:
Inclusion Criteria:

* Headache frequency of at least 1 per week for a minimum of 3 months
* Secondary Headache (cervical spine dysfunction)
* International Classification of headache Disorder:

  1. Pain localized in the neck and occiput, which can spread to other areas in the head, such as forehead, orbital region, temples, vertex, or ears, usually unilateral.
  2. Pain is precipitated or aggravated by specific neck movements or sustained postures.
  3. At least one of the following:

     1. Resistance to or limitation of passive neck movements
     2. Changes in neck muscle contour, texture, tone, or response to active and passive stretching and contraction
     3. Abnormal tenderness of neck musculature

Exclusion Criteria:

* Other types of headache
* Trigger points of upper cervical muscles
* Congenital conditions of cervical spine
* Cervical Disc herniation
* Fracture
* Cervical Artery disease
* Red flags of Thrust Joint Manipulation

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-04 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 12th Day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain.

SECONDARY OUTCOMES:
Pressure Pain Threshold (PPT) | 12th Day
  Changes from Baseline Pressure Pain Threshold (PPT) were taken with the help of algometer.
Headache Disability Index | 12th Day
  Scoring instructions: Yes = 4 points, Sometimes = 2, No = 0. Using this system, a total score of 10-28 is considered to indicate mild disability; 30-48 is moderate disability; 50-68 is severe disability; 72 or more is complete disability
Range of Motion(ROM) Cervical (Flexion) | 12th Day
  Changes from the baseline ROM range of motion of cervical spine flexion was taken with the help of inclinometer
ROM Cervical (Extension) | 12th Day
  Changes from the baseline ROM range of motion of cervical spine Extension was taken with the help of inclinometer
ROM Cervical (Side Bend) | 12th Day
  Changes from the baseline ROM range of motion of cervical spine Side bending was taken with the help of inclinometer
ROM Cervical Rotation | 12th Day
  Changes from the baseline ROM range of motion of cervical spine rotation was taken with the help of inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Dr Saira Waqqar, PP-DPT, MHPE, Principal Investigator — Riphah International University
Locations (1):
- Max health Rehabilitation Centre, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sjaastad O, Saunte C, Hovdahl H, Breivik H, Gronbaek E. "Cervicogenic" headache. An hypothesis. Cephalalgia. 1983 Dec;3(4):249-56. doi: 10.1046/j.1468-2982.1983.0304249.x. No abstract available. PMID 6640659
- [Background] Sjaastad O, Fredriksen TA, Pfaffenrath V. Cervicogenic headache: diagnostic criteria. The Cervicogenic Headache International Study Group. Headache. 1998 Jun;38(6):442-5. doi: 10.1046/j.1526-4610.1998.3806442.x. No abstract available. PMID 9664748
- [Background] Haldeman S, Dagenais S. Cervicogenic headaches: a critical review. Spine J. 2001 Jan-Feb;1(1):31-46. doi: 10.1016/s1529-9430(01)00024-9. PMID 14588366
- [Background] Lord SM, Barnsley L, Wallis BJ, Bogduk N. Third occipital nerve headache: a prevalence study. J Neurol Neurosurg Psychiatry. 1994 Oct;57(10):1187-90. doi: 10.1136/jnnp.57.10.1187. PMID 7931379
- [Background] Fleming R, Forsythe S, Cook C. Influential variables associated with outcomes in patients with cervicogenic headache. J Man Manip Ther. 2007;15(3):155-64. doi: 10.1179/106698107790819846. PMID 19066663
- [Background] Evers S. Comparison of cervicogenic headache with migraine. Cephalalgia. 2008 Jul;28 Suppl 1:16-7. doi: 10.1111/j.1468-2982.2008.01609.x. No abstract available. PMID 18494987
- [Background] Bogduk N, Govind J. Cervicogenic headache: an assessment of the evidence on clinical diagnosis, invasive tests, and treatment. Lancet Neurol. 2009 Oct;8(10):959-68. doi: 10.1016/S1474-4422(09)70209-1. PMID 19747657
- [Background] van Suijlekom JA, Weber WE, van Kleef M. Cervicogenic headache: techniques of diagnostic nerve blocks. Clin Exp Rheumatol. 2000 Mar-Apr;18(2 Suppl 19):S39-44. PMID 10824286
- [Background] Biondi DM. Cervicogenic headache: diagnostic evaluation and treatment strategies. Curr Pain Headache Rep. 2001 Aug;5(4):361-8. doi: 10.1007/s11916-001-0026-x. PMID 11403740
- [Background] Bogduk N. The neck and headaches. Neurol Clin. 2004 Feb;22(1):151-71, vii. doi: 10.1016/S0733-8619(03)00100-2. PMID 15062532
- [Background] Jull G, Barrett C, Magee R, Ho P. Further clinical clarification of the muscle dysfunction in cervical headache. Cephalalgia. 1999 Apr;19(3):179-85. doi: 10.1046/j.1468-2982.1999.1903179.x. PMID 10234466
- [Background] Mohamed AA, Shendy WS, Semary M, Mourad HS, Battecha KH, Soliman ES, Sayed SHE, Mohamed GI. Combined use of cervical headache snag and cervical snag half rotation techniques in the treatment of cervicogenic headache. J Phys Ther Sci. 2019 Apr;31(4):376-381. doi: 10.1589/jpts.31.376. Epub 2019 Apr 1. PMID 31037013
- [Background] Umar M, Naeem A, Badshah M, Zaidi S. A randomized control trial to review the effectiveness of cervical mobilization combined with stretching exercises in cervicogenic headache. J Public Health Biolo Sci. 2012;1(1):09-13.
- [Background] Jamil M, Janjua U. Comparison of cervicogenic headache between housewives and working women. Rawal Medical Journal. 2020 Jan;45(1):77-9.
- [Background] Umar M, Badshah M, Maryam M, Naeem A, Rehman L, Ahmed M. Prevalence Of Different Types Of Headache In Medical Students Of Rawalpindi & Islamabad. International Journal of Rehabilitation Sciences (IJRS). 2018 Mar 15;4(01):15-9.
- [Background] Coelho M, Ela N, Garvin A, Cox C, Sloan W, Palaima M, et al. The effectiveness of manipulation and mobilization on pain and disability in individuals with cervicogenic and tension-type headaches: a systematic review and meta-analysis. Physical Therapy Reviews. 2019;24(1-2):29-43
- [Background] Rani M, Kulandaivelan S, Bansal A, Pawalia A. Physical therapy intervention for cervicogenic headache: an overview of systematic reviews. European Journal of Physiotherapy. 2019:1-7
- [Background] Rasul HNU, Dustagir A, Malik AN. Role of Mobilization to Improve Cervicogenic Headache